CLINICAL TRIAL: NCT00028067
Title: A Phase III Study Comparing the Antiviral Efficacy and Safety of Atazanavir With Nelfinavir: Each in Combination With Dual Nucleoside Therapy in HIV-Infected Subjects Who Have Failed a Regimen Not Containing a Protease Inhibitor
Brief Title: A Comparison of Atazanavir and Nelfinavir, Each in Combination With 2 NRTIs, in Patients Who Have Failed Treatments Without a Protease Inhibitor
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Purpose: Treatment
Other Study IDs: 302F; AI424-037
Record Dates: First submitted 2001-12-10; First posted 2001-12-11 (Estimated); Last update posted 2011-05-04 (Estimated); Status verified 2011-04

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; HIV Protease Inhibitors; RNA, Viral; Reverse Transcriptase Inhibitors; Viral Load; BMS 232632
MeSH Terms: conditions — HIV Infections | interventions — Atazanavir Sulfate; Nelfinavir

INTERVENTIONS:
Drug: Atazanavir
Drug: Nelfinavir mesylate

SUMMARY:
The purpose of this study is to compare the atazanavir and nelfinavir (NFV) treatments in their ability to reduce viral load.

DETAILED DESCRIPTION:
In this double-blind, double-placebo, randomized, 2-arm study, atazanavir and NFV each are given in combination with 2 open-label nucleoside reverse transcriptase inhibitors (NRTIs) over 48 weeks. Patients assigned to atazanavir will receive placebo capsules which are identical in size and appearance to NFV. Patients assigned to NFV will receive placebo capsules which are identical in size and appearance to atazanavir. HIV levels are monitored.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Have a viral load of 1000 or more copies/ml within 3 weeks before randomization. Have a CD4 cell count of 50 or more cells/mm3 within 3 weeks prior to randomization.
* Are at least 16 years old (or the minimum age by local requirements).
* Have had more than 16 weeks of therapy with a non-nucleoside reverse transcriptase inhibitor (NNRTI) and/or nucleoside reverse transcriptase inhibitor (NRTI).
* Use effective barrier method of contraception.
* Give written informed consent.
* Are available for follow-up for at least 52 weeks.

Exclusion Criteria

Patients may not be eligible for this study if they:

* Have used a protease inhibitor (PI) treatment for more than 7 days or within 30 days prior to screening.
* Have a newly-diagnosed HIV-related infection or any medical condition requiring relatively short but intense therapy at the time of enrollment.
* Have hepatitis in the 30 days before the study. Patients with long-term hepatitis are eligible if their liver function meets certain requirements.
* Are unable to demonstrate responsiveness to a provided NRTI.
* Have had previous or expect a need for therapy with agents that may cause damage to nerve tissue, the pancreas, the liver, bone marrow, or cells within 3 months of study start.
* Use too much alcohol or drugs to be able to follow the study therapy; or if they use enough to increase the risk of developing pancreatitis or chemical hepatitis.
* Have severe diarrhea within 30 days prior to study entry.
* Are pregnant or breast-feeding.
* Have a history of hemophilia.
* Have history or signs of bilateral peripheral neuropathy.
* Have cardiomyopathy.
* Have certain heart problems.
* Cannot tolerate oral medication.
* Have any other problems that would interfere with the study.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500
Dates: Start 2001-08; Primary Completion 2002-04 (Actual); Study Completion 2002-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Giordano, Study Director
Locations (62):
- United States (47):
  - Health for Life Clinic, Little Rock, Arkansas
  - East Bay AIDS Ctr, Berkeley, California
  - Orange County Ctr for Special Immunology, Fountain Valley, California
  - Tower Infectious Diseases, Los Angeles, California
  - Kaiser Hospital, Sacramento, California
  - HIV Institute / Davies Med Ctr, San Francisco, California
  - Kaiser Foundation Hospital, San Francisco, California
  - IDC Research Initiative, Altamonte Springs, Florida
  - Larry Bush, Atlantis, Florida
  - Bach and Godofsky, Bradenton, Florida
  - North Broward Hosp District / HIV Clinical Research, Fort Lauderdale, Florida
  - Gary Richmond MD, Fort Lauderdale, Florida
  - Infectious Diseases Associates, Sarasota, Florida
  - Daniel Seekins, Tampa, Florida
  - Infectious Disease Research Inst, Tampa, Florida
  - Philip Brachman, Atlanta, Georgia
  - Med College of Georgia, Augusta, Georgia
  - Cook County Gen Hosp / Division of Infect Diseases, Chicago, Illinois
  - Division of Inf Diseases/ Indiana Univ Hosp, Indianapolis, Indiana
  - Tulane Univ School of Medicine, New Orleans, Louisiana
  - Beth Israel Deaconess Med Ctr, Boston, Massachusetts
  - Community Research Initiative of New England, Brookline, Massachusetts
  - CRI - Springfield, Springfield, Massachusetts
  - Henry Ford Hosp, Detroit, Michigan
  - Infectious Disease Clinic, Warren, Michigan
  - Washington Univ School of Medicine, St Louis, Missouri
  - South Jersey Infectious Diseases Inc, Somers Point, New Jersey
  - Community Research Initiative on AIDS, New York, New York
  - Saint Luke's - Roosevelt Hosp Ctr, New York, New York
  - Mount Sinai Med Ctr, New York, New York
  - Albert Einstein College of Medicine, The Bronx, New York
  - Carolinas Med Ctr, Charlotte, North Carolina
  - Piedmont Infectious Disease Consultants, Hickory, North Carolina
  - Jemsek Clinic, Huntersville, North Carolina
  - Wake Forest Univ School of Medicine, Winston-Salem, North Carolina
  - Summa Health System, Akron, Ohio
  - Associates in Med and Mental Health, Tulsa, Oklahoma
  - Research & Education Group, Portland, Oregon
  - Hahnemann Univ Hosp, Philadelphia, Pennsylvania
  - Ludwig Lettau Private Practice, Charleston, South Carolina
  - Univ of South Carolina School of Medicine, Columbia, South Carolina
  - North Texas Center for AIDS & Clinical Research, Dallas, Texas
  - Univ of Texas Southwestern Med Ctr, Dallas, Texas
  - Joseph Gathe, Houston, Texas
  - Univ TX Health Science Ctr, Houston, Texas
  - Hampton Roads Med Specialists, Hampton, Virginia
  - Wisconsin AIDS Research Consortium, Milwaukee, Wisconsin
- Canada (5):
  - Downtown Infectious Diseases Clinic, Vancouver, British Columbia
  - McMaster Univ Med Ctr, Hamilton, Ontario
  - Sunnybrook Health Science Ctr, Toronto, Ontario
  - Clinique Medicale du Quartier Latin, Montreal, Quebec
  - Clinique Medicale L'Actuele, Montreal, Quebec
- Mexico (4):
  - Hospital General De Mexico, Mexico City
  - Hospital Regional, Mexico City
  - Instituto Nacional de Enfermedades Respiratorias, Mexico City
  - Instituto Nacional de la Nutricion, Mexico City
- Puerto Rico (2):
  - Ponce School of Medicine, Ponce
  - Hepatology / Infectious Diseases, Santruce
- Thailand (4):
  - Program on AIDS / Thai Red Cross Society, Bangkok
  - Ramathibodi Hosp, Bangkok
  - Siriraj Hosp / Mahidol Univ, Bangkok
  - Khonkaen Univ, Khonkaen